CLINICAL TRIAL: NCT02436928
Title: A Study to Evaluate the Safety and Immunogenicity of H7N9 Influenza Vaccine (AT-501) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-MV-21
Record Dates: First submitted 2015-04-27; First posted 2015-05-07 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-03

CONDITIONS: H7N9 Influenza Vaccine
Keywords: H7N9 Influenza; Avian influenza A; cell culture derived
MeSH Terms: interventions — Vaccines; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AT-501 High Dose vaccine (Experimental): Inactivated H7N9 High Dose Antigen
  Interventions: Biological: AT-501 High Dose vaccine
- AT-501 High Dose vaccine with Adjuvant (Experimental): Inactivated H7N9 High Dose Antigen with Adjuvant
  Interventions: Biological: AT-501 High Dose vaccine with Adjuvant
- AT-501 Low Dose vaccine (Experimental): Inactivated H7N9 Low Dose Antigen
  Interventions: Biological: AT-501 Low Dose vaccine
- AT-501 Low Dose vaccine with Adjuvant (Experimental): Inactivated H7N9 Low Dose Antigen with Adjuvant
  Interventions: Biological: AT-501 Low Dose vaccine with Adjuvant

INTERVENTIONS:
Biological: AT-501 High Dose vaccine — Comparison of each dose of vaccine
  Arms: AT-501 High Dose vaccine
Biological: AT-501 High Dose vaccine with Adjuvant — Comparison of each dose of vaccine
  Arms: AT-501 High Dose vaccine with Adjuvant
Biological: AT-501 Low Dose vaccine — Comparison of each dose of vaccine
  Arms: AT-501 Low Dose vaccine
Biological: AT-501 Low Dose vaccine with Adjuvant — Comparison of each dose of vaccine
  Arms: AT-501 Low Dose vaccine with Adjuvant

SUMMARY:
This study aims to evaluate the safety and immunogenicity of an inactivated cell culture derived H7N9 vaccine in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject within the age limit range, is free of obvious health problems as judged by the investigator before entering the study.
2. Female subjects must be:

   * either of non-childbearing potential, or one year post-menopausal;
   * or, if of childbearing potential, must be abstinent or have used adequate contraceptive precautions for 30 days prior to receiving the study vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
3. Subject is willing and able to comply with all required study visits and follow-up required by this protocol.
4. Subject must provide written informed consent or the Subjects' legal representative must understand and consent to the procedure.

Exclusion Criteria:

1. Subjects with previous known or potential exposure to avian influenza virus H7N9 HA antigen and any other avian influenza including H5N1.
2. Subjects who have had seasonal influenza vaccine within 6 months prior to enrolment or who will have seasonal influenza vaccine at any time during the study period
3. Subjects administered with any other vaccine during the period within 6 weeks before the first administration of study vaccine.
4. Subjects with confirmed or suspected abnormal immune function, immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
5. Subjects with a history of hypersensitivity to vaccines or a history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
6. Subjects with a history of inflammatory or degenerative neurological disease .
7. Subjects receiving chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. Inhaled and topical steroids are allowed.
8. Known HIV, hepatitis B (HBsAg) or hepatitis C seropositivity.
9. Subjects, judged by the investigator, with any clinically significant medical illness including acute pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history, physical examination and/or laboratory screening tests.
10. The subjects would not be suitable for the vaccination if the screening laboratory tests show any of the follows

    * ALT or AST > upper limit of normal range (ULN);
    * Serum creatinine > upper limit of normal range (ULN);
    * Any significant laboratory abnormality as judged by the investigator
11. Subjects receiving administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or at any time during the study.
12. Subjects with acute disease at the time of enrolment.
13. Use of any investigational or non-registered product other than the study vaccine within 30 days prior to the first vaccination, or planned use of the abovementioned product during the entire study period.
14. Psychiatric, addictive, or any disorder, which may compromise the ability to give a truly informed consent for participation of this study or adequate compliance.
15. Any clinically relevant disease and/or abnormal laboratory findings (, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study.
16. Breast feeding or pregnant women or refusal to submit to a urine test to rule out pregnancy prior to enrolment and during the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety of AT-501 vaccine measured by Adverse Event | 1 year from the start of study enrolment
  Phase 1
  * Percentage, intensity and relationship to vaccination of solicited local and general signs and symptoms during a 7-day follow-up period after the first and second dose of administered vaccine.
  * Percentage, intensity and relationship to vaccination of unsolicited local and general signs and symptoms during a 21-day follow-up period after each administered vaccine.
  * Occurrence of overall adverse events and serious adverse events during the entire period of study.
Immunogenicity of AT-501 vaccine measured by HI titers | 1 year from the start of study enrolment
  Phase 2
  HI titers as follows:
  * Seroconversion Rate (SCR) at day 22 and 43
  * Seroconversion Factor (SCF) at day 22 and day 43
  * Seroprotection Rate (SPR) at day 22 and day 43

SECONDARY OUTCOMES:
Immunogenicity of AT-501 vaccine measured HI and neutralizing antibody titers | 1 year from the start of study enrolment
  Phase 1
  * Change of antibody titers from baseline to day 22 and day 43
  * Geometric Mean Titer (GMT) of both serum HI titers and neutralizing antibody titers, pre-vaccination and day 22 and day 43 post-vaccination
Safety of AT-501 vaccine measured by Adverse Event | 1 year from the start of study enrolment
  Phase 2
  * Percentage, intensity and relationship to vaccination of solicited local and general signs and symptoms during a 7-day follow-up period after the first and second dose of administered vaccine.
  * Percentage, intensity and relationship to vaccination of unsolicited local and general signs and symptoms during a 21-day follow-up period after each administered vaccine.
  * Occurrence of overall adverse events and serious adverse events during the entire period of study.

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Chwen Chang, Dr., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu UI, Hsieh SM, Lee WS, Wang NC, Kung HC, Ou TY, Chen FL, Lin TY, Chen YC, Chang SC. Safety and immunogenicity of an inactivated cell culture-derived H7N9 influenza vaccine in healthy adults: A phase I/II, prospective, randomized, open-label trial. Vaccine. 2017 Jul 24;35(33):4099-4104. doi: 10.1016/j.vaccine.2017.06.044. Epub 2017 Jun 28. PMID 28668573